CLINICAL TRIAL: NCT00006451
Title: T-cell Depletion In Unrelated Donor Marrow Transplantation
Brief Title: Bone Marrow Transplantation in Treating Patients With Leukemia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated (due to no accrual)
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: John Wagner, M.D., Masonic Cancer Center, University of Minnesota
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 1996LS142; UMN-MT-9506 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2000-11-06; First posted 2004-06-09 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2017-11

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma
Keywords: recurrent childhood acute lymphoblastic leukemia; stage IV childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; acute undifferentiated leukemia; stage IV adult lymphoblastic lymphoma; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; Methotrexate; Methylprednisolone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Procedure: radiation therapy

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill cancer cells.

PURPOSE: Randomized phase II/III trial to determine the effectiveness of bone marrow transplantation in treating patients who have leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare unrelated donor bone marrow transplantation using T-cell-depleted marrow versus unmodified marrow in adults and children with leukemia. II. Evaluate 2-year leukemia-free survival, primary and secondary graft failure, graft-versus-host disease, infection, and relapse in these patients. III. Assess the quality of life associated with T-cell-depleted versus unmodified, unrelated donor transplantation.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center. Patients receive myeloablative therapy according to diagnosis: those with acute lymphocytic leukemia and lymphoblastic lymphoma are treated with total body irradiation (TBI), with a testicular and chest wall boost as appropriate, followed by cyclophosphamide (CTX); patients with undifferentiated or biphenotypic leukemia or with acute or chronic myelocytic leukemia are treated with CTX followed by TBI. Patients are then randomly assigned to receive non-T-cell-depleted, unrelated marrow versus T-cell-depleted, unrelated marrow. The modified marrow is depleted of T-lymphocytes by counterflow elutriation and positively selected for CD34 cells. Graft-versus-host disease (GVHD) prophylaxis with cyclosporine and methotrexate is given to the unmodified marrow group. Patients who receive modified marrow are given antithymocyte globulin (or methylprednisolone) for graft rejection prophylaxis before transplantation and cyclosporine and methylprednisolone for GVHD prophylaxis after transplantation.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myelocytic leukemia with or without history of myelodysplastic syndrome Not in first complete remission (i.e., greater than 5% blasts in marrow) with t(8;21), t(15;17), or 16q abnormality unless failure on first-line induction therapy Acute lymphocytic leukemia (ALL) in one of the following categories: In second or third complete remission (CR) High-risk ALL in first CR, with high risk defined as: Hypodiploidy OR pseudodiploidy with t(9;22), t(4;11), or t(8;14) Failure to achieve CR after 4 weeks of induction therapy Elevated WBC at presentation, i.e.: Greater than 100,000 in patients aged 6 to 12 months Greater than 200,000 in patients aged 1 to 20 years Greater than 20,000 in patients aged 21 to 44 years Chronic myelogenous leukemia not in blast crisis (i.e., no greater than 30% promyelocytes plus blasts in bone marrow) Stage IV lymphoblastic lymphoma Undifferentiated or biphenotypic leukemia Unrelated donor available Patients aged 35 and younger: HLA-A, and -B serologic identity and HLA-DRB1 identity by high-resolution DNA typing OR Single HLA-A or -B serologic mismatch with DRB1 identity by high-resolution DNA typing OR HLA-A and -B serologic identity with single DRB1 mismatch by high- or low- resolution DNA typing Patients aged 36 to 44: HLA-A and -B serologic identity and HLA-DRB1 identity by high-resolution DNA typing The following exclude: Relapse 12 months after discontinuing therapy in patients aged 1 to 10 years who are in second remission Active central nervous system or leukemic skin involvement Requirement for additional mediastinal irradiation

PATIENT CHARACTERISTICS: Age: Under 46 Performance status: Karnofsky 70-100% Lansky 50-100% Hematopoietic: See Disease Characteristics Hepatic: Bilirubin less than 2.5 mg/dL AST less than 3 times normal Renal: Creatinine normal OR Creatinine clearance greater than 60 mL/min Cardiovascular: Asymptomatic OR Resting LVEF greater than 40% and improves with exercise Pulmonary: Asymptomatic OR DLCO greater than 45% of predicted (corrected for hemoglobin) Other: HIV negative No uncontrolled viral, bacterial, or fungal infection Not pregnant or nursing

PRIOR CONCURRENT THERAPY: No prior bone marrow transplantation No prior radiotherapy that precludes total body irradiation

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 1996-04; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Wagner, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States